CLINICAL TRIAL: NCT00094315
Title: Cocaine Relapse Prevention II
Brief Title: Development of Human Laboratory Study Model of Cocaine Relapse Prevention II - 1
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Other Study IDs: NIDA-CTO-0014-1
Record Dates: First submitted 2004-10-15; First posted 2004-10-15 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2005-09

CONDITIONS: Cocaine-Related Disorders
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Cocaine

INTERVENTIONS:
Drug: Cocaine (IV)

SUMMARY:
To study of classical conditioning mechanisms associated with arousal, craving and cocaine use.

DETAILED DESCRIPTION:
This is a single-site, double-blind, placebo-controlled crossover study of classical conditioning mechanisms associated with arousal, craving and cocaine use.

ELIGIBILITY:
Inclusion Criteria:

* Be English-speaking volunteers who are cocaine dependent
* Be non-treatment seeking at the time of the study
* Meet DSM-IV criteria for cocaine dependence
* Have ECG showing normal sinus rhythm, normal conductivity, and non clinically significant arrhythmias
* Females must provide a negative pregnancy test and agree to use birth control
* Have baseline laboratory tests within normal limits

Exclusion Criteria:

* Please contact site for more information

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16
Dates: Start 2004-09; Study Completion 2005-07

PRIMARY OUTCOMES:
Stimulated and non-stimulated craving
Cocaine assessment

CONTACTS AND LOCATIONS:
Overall Officials: John Roache, Ph.D., Principal Investigator — University of Texas
Locations (1):
- University of Texas Health Science Center, San Antonio, Texas, United States